CLINICAL TRIAL: NCT06101342
Title: A Phase 2, Open-Label, Multicenter, Randomized Study to Evaluate the Pharmacokinetics and Safety of Twice Yearly Long-Acting Subcutaneous Lenacapavir for Pre-Exposure Prophylaxis in People Who Inject Drugs
Brief Title: Study of Lenacapavir and Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF) for Prevention of HIV in People Who Inject Drugs (HPTN 103)
Acronym: PURPOSE 4
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: HIV Prevention Trials Network (Network); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GS-US-528-6363
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Pre-Exposure Prophylaxis of HIV Infection
MeSH Terms: interventions — lenacapavir; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Randomized Phase: Lenacapavir (LEN) Group (Experimental): Participants will receive subcutaneous (SC) LEN 927 mg on Day 1 and Week 26 and oral LEN 600 mg on Days 1 and 2.
  Interventions: Drug: Lenacapavir Injection; Drug: Lenacapavir Tablet
- Randomized Phase: Emtricitabine/ Tenofovir Disoproxil Fumarate (F/TDF) Group (Experimental): Participants will receive daily F/TDF (200/300 mg) fixed dose combination (FDC) tablets for up to 52 weeks.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate (F/TDF)
- Open-label Extension Phase: LEN (Experimental): Participants randomized to LEN in the Randomized Phase who choose to participate in the LEN Open-Label Extension (OLE) Phase will receive SC LEN every 26 weeks (± 7 days) and have study visits every 13 weeks (± 7 days). Participants randomized to F/TDF in the Randomized Phase who choose to participate in LEN OLE Phase will switch to SC LEN and have study visits at LEN OLE Day 1, Week 4 (± 2 days), Week 13 (± 7 days), and every 13 weeks (± 7 days) thereafter. SC LEN will be administered at the LEN OLE Day 1 visit and every 26 weeks thereafter. These participants will also receive loading doses of oral LEN on OLE Days 1 and 2. Upon completion of the LEN OLE Phase, participants will transition to local HIV prevention services and return for a 30-day follow-up visit. At that time, participation in the study will end.
  Interventions: Drug: Lenacapavir Injection; Drug: Lenacapavir Tablet
- Pharmacokinetic (PK) Tail Phase: F/TDF (Experimental): Participants eligible for the PK Tail Phase will receive open-label oral F/TDF once daily for up to 78 weeks and complete study visits every 13 weeks (± 7 days). PK Tail Day 1 visit will occur 26 weeks (± 7 days) after the last SC LEN injection.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate (F/TDF)

INTERVENTIONS:
Drug: Lenacapavir Injection — Administered subcutaneously
  Other Names: GS-6207; Yeztugo®
  Arms: Open-label Extension Phase: LEN; Randomized Phase: Lenacapavir (LEN) Group
Drug: Lenacapavir Tablet — Administered orally
  Other Names: GS-6207
  Arms: Open-label Extension Phase: LEN; Randomized Phase: Lenacapavir (LEN) Group
Drug: Emtricitabine/tenofovir disoproxil fumarate (F/TDF) — Administered orally
  Other Names: Truvada®
  Arms: Pharmacokinetic (PK) Tail Phase: F/TDF; Randomized Phase: Emtricitabine/ Tenofovir Disoproxil Fumarate (F/TDF) Group

SUMMARY:
The goals of this clinical study are to look at how lenacapavir (LEN) passes through the body and to assess the safety of LEN and emtricitabine/tenofovir disoproxil fumarate (F/TDF) for pre-exposure prophylaxis (PrEP) in people who inject drugs (PWID) in the United States (US).

The primary objectives of this study are to characterize the pharmacokinetics (PK) of LEN and to evaluate the safety of LEN and F/TDF for PrEP in US PWID.

ELIGIBILITY:
Key Inclusion Criteria:

* Urine drug screen positive for any drug of misuse including, but not limited to, opioids (eg, fentanyl, heroin), stimulants (eg, cocaine, amphetamines), psychoactive drugs (eg, benzodiazepines), or a combination of these drugs.
* Evidence of recent injection (eg, track marks).
* Self-report of injection paraphernalia sharing in the prior 30 days.
* Hepatitis B virus (HBV) surface antigen (HBsAg) negative.
* Negative local rapid HIV-1/2 antibody (Ab)/antigen (Ag) test, central HIV-1/2 Ab/Ag, and HIV-1 RNA quantitative nucleic acid amplification testing (NAAT).
* Estimated glomerular filtration rate (GFR) at least 60 mL/min at screening according to the Cockcroft-Gault formula for creatinine clearance (CLcr).

Key Exclusion Criteria:

* Self-reported history of previous positive results on an HIV test.
* Any reactive or positive HIV test result at screening or enrollment, even if HIV infection is not confirmed.
* Coenrollment in any other interventional research study or other concurrent studies that may interfere with this study (as provided by self-report or other available documentation) without prior approval from the Medical Monitor/Joint Clinical Management Committee while participating in this study.
* Past or current participation in HIV vaccine or HIV broadly neutralizing antibody study unless individual provides documentation of receipt of placebo (ie, not active product).
* Prior use of long-acting systemic pre-exposure prophylaxis (PrEP) (including cabotegravir (CAB) or islatravir studies).
* Acute viral hepatitis A or acute or chronic hepatitis B or C infection.
* Have a suspected or known active, serious infection(s) (eg, active tuberculosis, etc).
* Evidence of moderate or severe liver fibrosis or a history of or current clinical decompensated liver cirrhosis (eg, ascites, encephalopathy, variceal bleeding). In individuals with active hepatitis C, Fibrosis-4 (FIB-4) score > 3.25 (formula provided below).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Ctrough for Lenacapavir (LEN): LEN Plasma concentration at the End of the Dosing Interval (Week 26) | Week 26
PK Parameter: Ctrough for LEN: LEN Plasma concentration at the End of the Dosing Interval (Week 52) | Week 52
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 30 days post last dose at Week 78
Percentage of Participants Experiencing Treatment-emergent Clinical Laboratory Abnormalities with LEN and F/TDF | First dose date up to 30 days post last dose at Week 78

SECONDARY OUTCOMES:
General Acceptability of LEN and F/TDF as PrEP as Assessed by Percentage of Participants with Acceptability Questionnaire Responses | Up to Week 52
  To assess the acceptability of the study drug, the participants will complete questionnaire including a question on general acceptability of the assigned study drug on an ordinal 5-category scale with a response of: Completely unacceptable, Unacceptable, No opinion, Acceptable, or Completely acceptable.
Satisfaction With Use of LEN and F/TDF as PrEP as Assessed by Percentage of Participants with Satisfaction Questionnaire Responses | Up to Week 52
  To assess the satisfaction with use of the study drug, the participants will complete questionnaire including a question on satisfaction with use of the assigned study drug on an ordinal 5-category scale with a response of: Very satisfied, Satisfied, Neutral, Dissatisfied, or Very dissatisfied.
Willingness to Use LEN and F/TDF as PrEP as Assessed by Percentage of Participants with Willingness to Use Questionnaire Responses | Up to Week 52
  To assess the willingness to use the study drug, the participants will complete questionnaire including a question on willingness to use the assigned study drug on an ordinal 5-category scale with a response of: Definitely Yes, Probably yes, Not sure/undecided, Probably No, or Definitely No.
Number of Participants with Adherence to LEN, as Assessed by On-time LEN Injections Received | Up to Week 26
Number of Participants with Adherence to F/TDF as Assessed by Adherence Levels Based on Intracellular Tenofovir-diphosphate (TFV-DP) Concentrations in Dried Blood Spot (DBS) | Up to Week 78

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (9):
- United States (9):
  - UCLA Vine Street Clinic, Los Angeles, California
  - UCSD AntiViral Research Center (AVRC), San Diego, California
  - University of Miami - Converge Miami Building, Miami, Florida
  - Johns Hopkins Medicine Institute for Clinical and Translational Research, Clinical Research, Baltimore, Maryland
  - Rutgers New Jersey Medical School, Department of Medicine, Newark, New Jersey
  - ICAP at Columbia University- Bronx Prevention Center, The Bronx, New York
  - University of Pennsylvania, Division of Infectious Diseases Penn Prevention Research Unit, Philadelphia, Pennsylvania
  - Houston AIDS Research Team CRS, Houston, Texas
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez S, Garcia-Romeu A, Wisdom J, Jones J. Methamphetamine use and HIV prevention: a qualitative study on challenges and opportunities for PrEP utilization. AIDS Care. 2026 Jan 7:1-14. doi: 10.1080/09540121.2025.2611079. Online ahead of print. PMID 41498432
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06101342